CLINICAL TRIAL: NCT06451172
Title: Novel Antisense Oligonucleotide Eye Drops for Treating Antibiotic-Resistant Bacterial Keratitis
Acronym: ASOTARI
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202301V1; Fudan Eye and ENT Hospital (Other: 202301V1)
Record Dates: First submitted 2024-05-28; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Bacterial Keratitis; Antibiotic-resistant Bacteria; Infections, Bacterial; Corneal Diseases; Eye Diseases; Vision Disorders; Sensation Disorders; Blindness; Antisense Peptide Nucleic Acid; Antibacterial Therapy
Keywords: Bacterial Keratitis; Infections, Bacterial; Corneal Diseases; Eye Diseases
MeSH Terms: conditions — Bacterial Infections; Corneal Diseases; Eye Diseases; Vision Disorders; Sensation Disorders; Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASO Single Group (Experimental): ASO eye drops are used through the local administration. Dosage form: eye drop solution. Dose:20uL. Frequency of administration: 3 times per day.
  Interventions: Drug: ASO

INTERVENTIONS:
Drug: ASO — Anticipated 20 Participants will receive a single group administered via eye drops in the study eye.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of GP-asPNA for in vivo treatment of severe antibiotic resistant bacterial keratitis.

DETAILED DESCRIPTION:
This is a study of antisense oligonucleotides (ASOs) in adult (ages 18 to 70) participants with severe antibiotic resistant bacterial keratitis. Approximately 20 participants will be enrolled.

Infectious keratitis or endophthalmitis, mainly caused by the trauma or intraocular surgical operation, has posed a grave threat to human vision health. Among them, infectious keratitis is the most common blinding keratopathy in developing countries. We develop a novel kind of Trojan strategy to specifically deliver ASOs into diverse bacteria rather than mammalian cells through the bacterial-specific ATP-binding cassette (ABC) sugar transporter. Compared with their cell-penetrating peptide counterparts, the antisense peptide nucleic acid modified with glucose polymer can be selectively internalized into human-derived multidrug- resistant Escherichia coli and methicillin-resistant Staphylococcus aureus, and they display a much higher uptake rate.

The follow-up period was 90 days, and the patients will be followed up 1 days, 3±1 days, 7±1 days, 14±2 days, 30±2 days, and 90±5 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* The results of antimicrobial susceptibility testing in patients with bacterial keratitis showed multidrug-resistant bacterial infections, and the existing commercial antibiotics could not effectively control the disease.
* Age over 18 years.
* No systemic immune eye disease.
* Good eyelid structure and blink function.
* Exists the potential of visual recovery by evaluation of ocular structure and function.
* Subjects or their legal guardians voluntarily participate in this study, sign informed consent, good compliance and cooperation with follow-up visits.

Exclusion Criteria:

* Lacrimal coating and blink function loss.
* Schirmer's test result is less than 2mm for severe dry eye disease.
* Pregnant and lactating women (pregnancy defined in this study as positive urine pregnancy test).
* Currently is involved in clinical trials of other drugs or medical devices.
* Active eye infection (including but not limited to: blepharitis, infectious conjunctivitis, sclerotitis, endophthalmitis) in target eye or contralateral eye within 30 days prior to enrollment.
* Ocular surface malignant tumor.
* A history of allergic reaction or allergy to sodium luciferin, allergy to protein products used for treatment or diagnosis, allergy to ≥ 2 drugs or non-drug factors, or current allergic disease.
* current in an infectious disease requiring oral, intramuscular or intravenous administration.
* Patients with systemic immune diseases.
* Any uncontrolled clinical problems (such as severe mental, neurological, cardiovascular, respiratory and other systemic diseases and malignant neoplasms).
* Not effective contraception.
* In uncontrolled hypertension, systolic is no less than 160 mmhg, diastolic is no less than 100 mmhg.
* In uncontrolled diabetes, fasting glucose is no less than 10.0umol/L.
* Renal insufficiency, serum creatinine is more than 133umol/L.
* Arrhythmia, myocardial ischemia, myocardial infarction (diagnosed by electrocardiogram).
* Liver dysfunction, al ANINE aminotransferase and aspartate aminotransferase levels are higher than 80 IU/L.
* Platelet level is below 100,000 /uL or above 450,000 /uL.
* Hemoglobin level is below 10.0g/dL (male) or 9.0g/dL (female).
* No anticoagulant was used, prothrombin time is higher than 16s, and thrombin time of activated part is higher than 50s.
* HIV infection (HIV-positive).
* Subjects lack compliance with the study or the ability to sign informed consent.
* There are currently signs of systemic infection, including fever and ongoing antibiotic treatment (in this study, systemic infection was defined as deviation from normal values of white blood cells, lymphocytes, and neutrophils on routine blood tests).
* Administration of Glucocorticoids and other systemic immunosuppressive drugs.
* The investigator judges other conditions unsuitable for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Bacteria testing outcome of the intervention eye | 90 Days
  Assess the efficacy of bacteria clearance based on RNA sequencing data using techniques such as ELISA and PCR. For instance, real-time polymerase chain reaction (PCR) is utilized to identify 16S rRNA in corneal biopsy samples.
Ophthalmic therapeutic effect of ASO eye drops | 90 Days
  Measure the decrease in size, depth and infiltrate of the ulcer in millimeters by slit lamp biomicroscopy.

SECONDARY OUTCOMES:
Visual improvement compared with baseline | 90 Days
  Judge the visual recovery progress according to visual examination results on day 1，3±1，7±1，14±2，30±2，90±5.

CONTACTS AND LOCATIONS:
Overall Officials: Jiaxu Hong, M.D., Ph.D, Study Director — Eye, and ENT Hospital,Shanghai Medical College, Fudan University,Shanghai, China
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Austin A, Lietman T, Rose-Nussbaumer J. Update on the Management of Infectious Keratitis. Ophthalmology. 2017 Nov;124(11):1678-1689. doi: 10.1016/j.ophtha.2017.05.012. Epub 2017 Sep 21. PMID 28942073
- [Result] Brown ED, Wright GD. Antibacterial drug discovery in the resistance era. Nature. 2016 Jan 21;529(7586):336-43. doi: 10.1038/nature17042. PMID 26791724
- [Result] Liu M, Chu B, Sun R, Ding J, Ye H, Yang Y, Wu Y, Shi H, Song B, He Y, Wang H, Hong J. Antisense Oligonucleotides Selectively Enter Human-Derived Antibiotic-Resistant Bacteria through Bacterial-Specific ATP-Binding Cassette Sugar Transporter. Adv Mater. 2023 Jul;35(28):e2300477. doi: 10.1002/adma.202300477. Epub 2023 May 26. PMID 37002615
- [Result] Zhang Q, Song B, Xu Y, Yang Y, Ji J, Cao W, Lu J, Ding J, Cao H, Chu B, Hong J, Wang H, He Y. In vivo bioluminescence imaging of natural bacteria within deep tissues via ATP-binding cassette sugar transporter. Nat Commun. 2023 Apr 22;14(1):2331. doi: 10.1038/s41467-023-37827-9. PMID 37087540